CLINICAL TRIAL: NCT05323825
Title: Randomized, Double-blind, Clinical Trial to Evaluate the Effect of a Fermented Dairy Food With Probiotics on Mental Performance
Brief Title: Effect of a Fermented Dairy Food With Probiotics on Mental Performance
Acronym: ShotRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00026
Record Dates: First submitted 2022-03-26; First posted 2022-04-12 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Change
Keywords: Probiotic; Fermented milk
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The content of the package is 100 g and should be consumed once a day for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Control group (Placebo Comparator): The content of the package is 100 g and should be consumed once a day for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Fermented milk product containing a probiotic
  Arms: Experimental group
Dietary Supplement: Placebo — Product with identical characteristics to the experimental product.
  Arms: Control group

SUMMARY:
Single-center, randomized, double-blind, placebo-controlled clinical study with two study groups.

One group will consume a product with functional ingredients and the other group will consume a placebo product. will consume a placebo product.

DETAILED DESCRIPTION:
When individuals are included in the study they will be randomized in equal proportion to one of the 2 groups of the study. The randomization will be stratified by age taking into account 2 strata (1:1). The first stratum corresponds to an age range of 18 to 40 years and the second stratum to an age range of 41 to 60 years.

The subject must consume the product for 8 weeks and will have a visit 4 weeks later as a follow-up of the study.

At the visits the subject will perform a series of cognitive tests and the intestinal microbiota will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-60 years.
* Individuals with a diagnosis of mild-moderate stress according to the Cohen's perceived stress scale perceived stress scale (PSS-10).
* Subjects with poor adherence to the Mediterranean diet according to the PREDIMED questionnaire (value below 9 points)*.
* BMI between 19 and 30 kg/m2.

Exclusion Criteria:

* Present chronic and/or acute digestive pathologies that may interfere in the absorption of nutrients (inflammatory intestinal diseases, inflammatory bowel absorption of nutrients (inflammatory intestinal diseases, etc.), etc.)
* Intake of probiotics and/or prebiotics in the four weeks prior to the inclusion in the study.
* Individuals who are on antibiotic treatment or have completed an antibiotic treatment during the 30 days prior to inclusion in the study.
* Vegan diet.
* Being taking any type of supplementation that interacts with cognitive level in the 2 weeks prior to the start of the study.
* Individuals who had taken or were taking any medications or supplementation for stress management, mood, or to induce sleep in the 2 weeks prior to the start of the study.
* A history of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Consumption of 2 or more Standard Drink Units (UBE) daily or 17 weekly in women, or consume 4 or more UBE daily or 28 weekly in men.
* Smoking and non-smoking subjects who have modified their nicotinic habits in the last 3 months.
* Pregnant or lactating women.
* Been participating or have participated in another clinical trial in the 2 months prior to the study to the study.
* Unwillingness or inability to comply with the procedures of the clinical trial.
* Subjects with any diagnosed psychiatric disorder.
* Subjects whose condition makes them ineligible for the study in accordance with the criteria of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | Change in baseline cognitive performance after 8 weeks of consumption
  COMPASS cognitive test panel

SECONDARY OUTCOMES:
Perceived Stress Scale | Day 1, at 4 and 8 weeks later
  PSS-14 test
Mood profile | Day 1, at 4 and 8 weeks later
  POMS test
Depression, Anxiety and Stress | Day 1, at 4 and 8 weeks later
  DASS21 test
State of mind | Day 1, at 4 and 8 weeks later
  PANAS test
Stress status using VAS scale | Day 1, at 4 and 8 weeks later
  Stress status on the day of the visit
Sleep efficiency | It will be measured for 3 days, before starting the consumption of the product, after 30 days of consumption and at the end of consumption (60 days).
  Measured by accelerometry, with Actigraph wGT3X-BT
Sleep quality | Day 1, at 4 and 8 weeks later
  Pittsburgh test
Gut microbiota | Day 1, at 4, 8 and 12 weeks later
  Evaluated with stool sample
Adverse events | At 4 weeks, 8 and 12 weeks after consumption
  It will be evaluated at each of the visits and in the month of follow-up will be evaluated with a daily diary.
Concomitant medication | Day 1, at 4, 8 and 12 weeks later
  The change in the use of medications will be evaluated. It will be evaluated at each of the visits and in the month of follow-up will be evaluated with a daily diary.
Dietary survey | Day 1, at 4, 8 and 12 weeks later
  Three days will be evaluated (two weekdays and one weekend day).
Body weight | Day 1, at 8 weeks later
  Bioimpedance, in Kg. For this we will use a TANITA
Liver safety variables | It will be measured twice, once at baseline or at the end of the consumption after 8 weeks.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Román, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain